CLINICAL TRIAL: NCT02679326
Title: The Efficacy of Treating Plantar Fasciitis With Therapeutic Ultrasound
Brief Title: Plantar Fasciitis and Therapeutic Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 4/2015
Record Dates: First submitted 2016-02-07; First posted 2016-02-10 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-01

CONDITIONS: Plantar Fasciitis
Keywords: Therapeutic ultrasound, Treatment, Plantar fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Ultrasonic Therapy

STUDY DESIGN:
Intervention Model Description: Double blinded RCT
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Experimental): will receive stretching guidance and high level active Ultrasound
  Interventions: Device: Therapeutic ultrasound
- control group (Placebo Comparator): will receive stretching guidance and very low level of Ultrasound
  Interventions: Device: Therapeutic ultrasound

INTERVENTIONS:
Device: Therapeutic ultrasound

SUMMARY:
The purpose of this study is to determine whether Therapeutic Ultrasound is effective in the treatment of Plantar fasciitis (PF).

DETAILED DESCRIPTION:
Plantar fasciitis (PF) is the main cause of pain in the bottom of the heel. According to the American Physical Therapy Association guidelines since 2008, many treatments have been described to correct the problem, but there are very few high level randomized trials that proved them. Although not mentioned even in clinical treatment guidelines in PF, one of the most common conservative treatments for use, in general and Israel in particular, is a therapeutic ultrasound device. Despite this widespread use, there are very few research evidence which examining the effectiveness of this device for the treatment of PF. The purpose of this study is to evaluate the effect of therapeutic ultrasound versus sham ultrasound on pain, function and quality of life of patients with PF. Our hypothesis is that the use of ultrasound parameters that cause an increase in the target tissue heat (from 1.75 to 1 W/cm2, Continues intensity of 1 MHZ) will result in a significant improvement than placebo. To evaluate this hypothesis, we will do a prospective, controlled, randomized, double-blind interventional clinical study. The study population will include 60 patients, aged 18 or older, suffering from PF and meet inclusion criteria. Subjects will be divided randomly into study or control group, Both groups will receive stretching Instructions, when the study group will Receive active ultrasound and the control group will Receive sham ultrasound. Both groups will receive 8 treatments, twice a week.

ELIGIBILITY:
Inclusion Criteria:

* Worsening symptoms first steps in the morning or at the beginning of walking after sitting for long periods, and after long walking or standing.
* Pain at the bottom of the heel produced by weight bearing or local press.
* Pain level 3 or higher on NPRS at first steps in the morning.
* Tenderness, swelling, or both in the region of proximal plantar fascia and at medial plantar tuberosity of the calcaneous.
* Gradual development of pain at the bottom of the heel.

Exclusion Criteria:

* Peripheral neuropathy.
* Tarsal tunnel syndrome (TTS) \ Fat Pad Syndrome (FPS).
* Calcaneal cyst, Fracture or bone cancer.
* Osteo Arthritis (OA) of the foot fingers or Rheumatoid arthritis (RA).
* Foot surgery at the last year.
* Steroid injections at the last six months.
* Pregnancy.
* Foot infection or diabetic foot.
* Stress fractures of the heel.
* Unavailability in advance to participate in research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05-28 (Actual); Study Completion 2017-05-28 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) at morning | at morning after 4 weeks of treatment
  pain level at the heel at the first step in the morning.

SECONDARY OUTCOMES:
NPRS during the day | 1 day
  pain level during the day.
Foot & Ankle computerized adaptive test (CAT) | 2 & 4 weeks of treatment
  Questionnaire of quality of life
Algometric test | 4 weeks of treatment
  Average of 3 testing of Pressure on the medial tuberosity

CONTACTS AND LOCATIONS:
Overall Officials: Ron Ben-izhak, PHD, Principal Investigator — Maccabi Healthcare Services, Israel
Locations (1):
- Maccabee Health Services Physical therapy Clinic, Rehovot, Southern District, Israel